CLINICAL TRIAL: NCT00529464
Title: A Randomized Trial of Spectroscopy Versus Standard Care in Cervical Intraepithelial Neoplasia
Brief Title: Spectroscopy Versus Standard Care in Cervical Cancer Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Two participants enrolled, both inevaluable.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0582
Record Dates: First submitted 2007-09-12; First posted 2007-09-14 (Estimated); Results first posted 2010-12-08 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2012-12

CONDITIONS: Cervical Cancer
Keywords: Cervical Intraepithelial Neoplasia; Cervical Dysplasia; Cervical Cancer; Fluorescence Spectroscopy; Colposcopy; Loop Electrical Excision Procedure; LEEP
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia | interventions — Spectrometry, Fluorescence; Colposcopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Colposcopy (Experimental): Colposcopy - a direct magnified inspection of cervix
  Interventions: Procedure: Colposcopy
- Colposcopy + Fluorescence Spectroscopy (Experimental): Colposcopy - a direct magnified inspection of cervix + Fluorescence Spectroscopy - electromagnetic spectroscopy which analyzes fluorescence from a sample.
  Interventions: Procedure: Fluorescence Spectroscopy; Procedure: Colposcopy
- Colposcopy + LEEP Procedure (Experimental): Colposcopy - a direct magnified inspection of cervix + loop electrosurgical excision procedure (LEEP) - thin, low-voltage electrified wire loop to cuts out cervix abnormal tissue.
  Interventions: Procedure: Colposcopy; Procedure: LEEP Procedure

INTERVENTIONS:
Procedure: Fluorescence Spectroscopy — Pictures of the cervix will be taken before and after the application of acetic acid. A clean probe will be placed against the cervix that sends out light and reads how much light is absorbed by the tissue.
  Arms: Colposcopy + Fluorescence Spectroscopy
Procedure: Colposcopy — A standard colposcopy will be performed.
Procedure: LEEP Procedure — A small heated wire loop is used to remove a cone-shaped piece of abnormal tissue. Procedure is performed on the same day as the colposcopy exam.
  Other Names: Loop Electrical Excision Procedure
  Arms: Colposcopy + LEEP Procedure

SUMMARY:
Primary objectives

1. To conduct a randomized clinical trial of the emerging technology fluorescence and reflectance spectroscopy, comparing colposcopy to colposcopy + spectroscopy in the diagnostic setting, stratifying patients by outside Papanicolaou (Pap) smear of low grade and high grade squamous intraepithelial lesions, and to use multispectral digital colposcopy retrospectively.

   The number of clinically read referral Paps, clinically read UT MD Anderson Cancer Center (MDACC) Paps, quantitatively read Paps, quantitatively read biopsies, point probe fluorescence/reflectance spectroscopy, and the multi-spectral digital colposcopy image, that shows a possible cancer, High-grade Squamous Intraepithelial Lesion (HGSIL), Low-grade Squamous Intraepithelial Lesion (LGSIL), or changes less than LGSIL to colposcopically directed biopsies at the first visit, Loop Electrical Excision Procedure (LEEP) at the second visit if needed, repeat evaluations at 6, 12, and 18 months that have Paps, or Paps + Endocervical Curettage or sample of the cervical canal + possible biopsy, and at the 24 month visit when all patients will at minimum have a Pap and an Endocervical Curettage for certain, and a cervical biopsy if any colposcopic abnormality is present.
2. To see if optical spectroscopy using both the point probe and the multi-spectral device improves diagnosis by improving specificity over colposcopy alone.

   1. To study the number of colposcopically directed biopsies that show High-grade Squamous Intraepithelial or cancer.
   2. To study the number of LEEP specimens that show HGSIL or cancer.

DETAILED DESCRIPTION:
A colposcopy is an exam of the cervix, using a magnifying lens. Fluorescence spectroscopy uses a special light source to look for abnormal cells during the colposcopy.

If you agree to take part in this study, depending on your referral Pap smear diagnosis, you will be randomly assigned (as in the toss of a coin) to one of 3 groups. Participants in Group 1 will undergo a standard colposcopy. Participants in Group 2 will undergo a colposcopy plus fluorescence spectroscopy. If your referral Pap smear diagnosis is high-grade dysplasia (abnormal tissue), you may be assigned to Group 3. Participants in Group 3 will have a colposcopy exam and a loop electrical excision procedure (LEEP--a procedure where a small heated wire loop is used to remove a cone-shaped piece of abnormal tissue) on the same day.

At Visit 1, your complete medical history will be recorded. You will have a physical exam. You will have a colposcopy. You will have a pap smear, and cultures will be taken for gonorrhea and chlamydia. The bodily fluid samples for the cultures are collected by using a cotton swab or cytobrush (the same kind of brush used to collect cells for a Pap smear) to collect mucous from the canal of the cervix. Blood (about 6 teaspoons) may be drawn for syphilis, hepatitis, and Human Immunodeficiency Virus (HIV) tests. You may have a Human Papilloma Virus (HPV) test. The HPV test is performed in the same manner as the bodily fluid sample collection. Depending on which arm you are assigned to, you may have an endocervical curette (ECC) and cervical biopsies of abnormal areas. Before you begin the study, you should ask your study doctor whether or not you were assigned to the group that will be receiving the ECC and cervical biopsies. During the ECC, cells/tissue will be scraped from the cervical canal with an instrument which is made to only take cells/tissue from the surface of the cervical canal. A cervical biopsy is when a tiny piece of tissue from the outside surface of the cervix is removed. Women who are able to have children must have a negative urine pregnancy test. You will complete a behavioral risk-factor interview and questionnaire. The questionnaire should take about 10 minutes to complete.

If you are in Group 2, at each visit you will have a picture of the cervix before and after the application of acetic acid. You will also have a clean probe, the size of a pencil, placed against your cervix. The probe sends out light and reads how much light is absorbed by the tissue. The reading will show doctors and nurses the types of molecules present in the cells of the cervix. Two (2) to 3 measurements will be made. Each measurement takes about a minute.

All participants will have routine visits every 6 months for 2 years. If you miss your scheduled appointment, the next available appointment will be scheduled for you. At these visits, study data will be collected. You will have a colposcopy and Pap smear. You will have cervical biopsies taken and an ECC (if a high-grade lesion is seen). You will have another HPV test.

If at your 24- month appointment there is a lesion on your cervix that can be seen by colposcopy, you will be treated with a loop electrosurgical excision cone procedure. This is a procedure where a tiny heated wire is used to remove the lesion from your cervix. If there is no lesion on your cervix that can be seen by colposcopy, researchers will take 1 cervical biopsy and an endocervical curettage.

You will be taken off study if the disease gets worse. You will be considered off study after the 24-month visit.

This is an investigational study. The spectroscopy device has not been approved by the FDA. It is authorized for use in research only. About 360 women will take part in this multicenter study. Up to 120 women will be enrolled at UT MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older
* Non-pregnant
* Patients with abnormal smears with cervical intraepithelial neoplasia (both low grade squamous intraepithelial lesions and high grade squamous intraepithelial lesions equal to cervical intraepithelial neoplasia 1-3)

Exclusion Criteria:

* Patients who have had cytotoxic chemotherapy within 12-months prior to enrolling in this study, since the chemotherapy often induces change in the cervix.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen E. Rhodes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (2):
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - UT MD Anderson Cancer Center, Houston, Texas
- British Columbia Cancer Research Centre, Vancouver, British Columbia, Canada

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 11/08/06 through 05/01/08. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Two patients were recruited, both ineligible, with no research related procedures performed. Study terminated early due to low enrollment.
Groups:
- Colposcopy + LEEP: Colposcopy - a direct magnified inspection of cervix + loop electrosurgical excision procedure (LEEP) - thin, low-voltage electrified wire loop to cuts out cervix abnormal tissue.
Period: Overall Study
Arm/Group | Colposcopy | Colposcopy + Fluorescence Spectroscopy | Colposcopy + LEEP
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Colposcopy | Colposcopy + Fluorescence Spectroscopy | Colposcopy + LEEP | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years]
Sex: Female, Male [Count of Participants; unit: Participants]

OUTCOME MEASURES:

1. Primary Outcome: Number of Unnecessary Loop Electrosurgical Excision Procedures (LEEP)
Description: A LEEP is unnecessary if histological examination results in diagnosis of low grade squamous intraepithelial lesion or normal. Comparison of 3 arms (colposcopy to colposcopy + spectroscopy, colposcopy + LEEP Procedure) in the diagnostic setting, stratifying participants by outside Papanicolaou (Pap) smear of low grade and high grade squamous intraepithelial lesions, and to use multispectral digital colposcopy retrospectively, in identifying unnecessary LEEPs performed.
Time Frame: Up to 2 years
Population: The primary outcome measure could not be assessed because no subject received randomized treatment assignment. The study was terminated.
Arm/Group | Colposcopy | Colposcopy + Fluorescence Spectroscopy | Colposcopy + LEEP
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Clinical care begins at the start of the study and continues for 2 years.
Arm/Group | Colposcopy | Colposcopy + Fluorescence Spectroscopy | Colposcopy + LEEP
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
This study was terminated due to difficulty enrolling subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No